CLINICAL TRIAL: NCT05538559
Title: The Effectiveness of Carie Care, Chemomechanical Caries Removal Technique in Primary Teeth (Randomized Controlled Clinical Trial)
Brief Title: Carie Care, Chemomechanical Caries Removal Technique in Primary Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Caries Removal 2022
Record Dates: First submitted 2022-09-10; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Dental Caries; Primary Teeth
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental)
  Interventions: Other: Chemomechanical caries removal by Carie-Care
- Control (Active Comparator)
  Interventions: Other: Mechanical caries removal by Atraumatic Restorative Technique

INTERVENTIONS:
Other: Chemomechanical caries removal by Carie-Care — caries in primary teeth will be removed using Carie-Care™ the chemomechanical agent.
  Arms: Test
Other: Mechanical caries removal by Atraumatic Restorative Technique — caries in primary teeth will be removed using the mechanical caries removal by ART method.
  Arms: Control

SUMMARY:
Chemomechanical caries removal systems have emerged as a possible valuable alternative to conventional rotary caries removal techniques in pediatric patients. Carie-Care™ is an economically minimally invasive approach that selectively removes caries-infected tissue leaving the caries-affected tissue to conserve tooth structure

ELIGIBILITY:
Inclusion Criteria:

* Open carious lesions with a moderately deep dentin carious lesion(scores five or six, according to the International Caries Detection and Assessment System[ICDAS].
* The access of the carious lesion has to be large enough to allow the penetration of the excavator
* Children with behavior rating 3 or 4 according to the Frankl scale

Exclusion Criteria:

* Clinical or radiographic evidence of pulp, furcation, or periapical pathosis
* Proximal caries evidenced by bitewing x-ray

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Time taken for caries removal | Through procedure completion
  The time taken for the procedures will be measured from the beginning of caries removal procedure till the cavity is confirmed to be free of caries with the help of a stop watch and will be recorded in seconds.
Efficacy of caries removal | Through procedure completion
  Caries removal will be rated according to the scoring criteria that range between score zero where caries is removed completely to score 5 where caries is present at the base,walls and margins of the cavity
Child pain perception | Through procedure completion
  The type of response obtained for each observation was given a numerical value (score) like Score 1 (comfort), Score 2 (mild discomfort), Score 3 (moderately painful), and Score 4 (painful)
Child behavior | Through procedure completion
  Score 1: Definitely positive, Good rapport with the dentist, interested in the dental procedures, laughing and enjoying the situation.
  Score 2: Positive, Acceptance of treatment; at times cautious, willingness to comply with the dentist, at times with reservation but patient follows the dentist's directions cooperatively.
  Score 3:Negative, Reluctant to accept treatment; uncooperative, some evidence of negative attitude but not pronounced, i.e. /sullen, withdrawn.
  Score 4: Definitely negative, Refusal of treatment, crying forcefully, fearful or any other overt evidence of extreme negativism.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt